CLINICAL TRIAL: NCT03630302
Title: Intraoperative Investigation of a Directional Lead and Local Field Potentials for the Optimization of Stimulation Efficacy
Acronym: INVENT
Status: Completed | Type: Observational
Sponsor: Abbott Medical Devices (Industry)
Collaborators: Baylor College of Medicine (Other); University of Houston (Other)
Responsible Party: Sponsor
Other Study IDs: CRD_931 INVENT
Record Dates: First submitted 2018-08-09; First posted 2018-08-14 (Actual); Results first posted 2021-05-28 (Actual); Last update posted 2021-05-28 (Actual); Status verified 2021-05

CONDITIONS: Parkinson

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

INTERVENTIONS:
Device: DBS — Deep Brain Stimulation

SUMMARY:
The current study aims to explore the functional use of LFPs recorded intraoperatively for the optimization of a directional DBS lead programming

Aim-1: To determine whether intraoperative LFPs recorded from the segmented DBS electrode can predict the optimal stimulation parameters.

Aim-2: Compare the therapeutic window for stimulation delivered through directional and conventional leads and determine if the spatiospectral LFP patterns correlate with the presence of stimulation side effects.

DETAILED DESCRIPTION:
This is a feasibility study designed to evaluate the usefulness of intraoperative LFP recordings obtained from the implanted DBS lead to predict ideal stimulation parameters. Additionally this study will compare the therapeutic window for stimulation delivered through directional and conventional leads and determine if the spatiospectral LFP patterns correlate with the presence of stimulation side effects.

Approximately 15 subjects will be enrolled in this clinical investigation. The clinical investigation will be conducted at 2 centers in the USA.

Subjects participating in this clinical investigation will monitored during DBS implant procedure and programming. The expected duration of enrollment is 8 months. The total duration of the clinical investigation is expected to be 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-70 years
* Ability to provide informed consent
* Diagnosis of idiopathic Parkinson's disease, and DBS consensus team review supporting the placement of STN DBS.

Exclusion Criteria:

* Subject is not a surgical candidate;
* In the Investigator's opinion the subject unable to tolerate multiple programming sessions within a single setting;
* Subject unable to comply with the follow-up schedule

Ages: 18 Years to 70 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: In this study the investigators will explore the predictive capacity of LFPs recorded from STN. In total, 15 patients undergoing bilateral STN DBS will be enrolled for this investigation over a 1-year period. The current surgical case load at BCM supports this level of enrollment. The details of implantation procedures and blinded trial design are given in the following sections
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2018-07-12 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2020-01-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- CHI St. Luke's Health Baylor College of Medicine Med. Ctr., Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Groups:
- LFP Recording Patients: All patients underwent STN DBS implants. The DBS leads were programmed by clinicians at initial visit and symptoms re-evaluated at 3 month post-operative visit. Local field potentials (LFPs) were recorded from 9 patients during the surgery of DBS implants. Hardware issue prevented LFP recordings from 1 patient.
Period: Surgery
Arm/Group | LFP Recording Patients
Started | 10
Completed | 9
Not Completed | 1
Not completed — hardware issue prevented LFP recordings | 1
Period: 3 Month Visit
Arm/Group | LFP Recording Patients
Started | 9
Completed | 7
Not Completed | 2
Not completed — Adverse Event | 2
Period: Data Post Analyses
Arm/Group | LFP Recording Patients
Started | 7
Completed | 5
Not Completed | 2
Not completed — IRB issues prevented data from being analyzed and transferred | 2

BASELINE CHARACTERISTICS:
Groups:
- All Patients: All patients underwent STN DBS implants
Arm/Group | All Patients
Number analyzed (Participants) | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.3 (5.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 6
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
How long has the patient been diagnosed with PD [Mean (Standard Deviation); unit: years] | 8.95 (4.11)

OUTCOME MEASURES:

1. Primary Outcome: Number of DBS Leads With Clinical Programming at 3 Months That Were Consistent With Predictions Via LFP Features After DBS Implant Procedure
Description: From all DBS leads (2 per patient):
  Local field potentials (LFPs) were measured intraoperatively during DBS implant. Features such as beta band power (10-30Hz), high-frequency oscillation power (200-400Hz, HFO), as well as the cross frequency coupling between beta band power and HFO (CFC) were extracted from the LFP recordings from all electrodes. Electrodes with the most beta band power, most HFOs, and most CFC were documented.
  At 3 month post-op visit, the clinically programmed stimulation electrodes were documented, and were compared to the electrodes documented from the intraoperative LFP measures. Both matches in the exact contact and the row at which the contacts were in were documented and compared.
Time Frame: LFPs were analyzed after DBS implant procedure, clinical programming were done at 3 month followup
Population: patients who had both LFP data and clinical programming results, all patients have bilateral implants
Measure: Count of Units; unit: DBS leads
Units Other Than Participants: DBS leads
Groups:
- LFP Analyses From Patients With Bilateral Implants: all DBS leads from all patients that LFP analyses were performed on and clinical programming were obtained
Arm/Group | LFP Analyses From Patients With Bilateral Implants
Number analyzed (Participants) | 5
Number analyzed (DBS leads) | 10
DBS leads
  DBS leads that had clinical programming contact that matched highest beta-band power | 2
  DBS leads that had clinical programming row that matched highest beta-band power | 3
  DBS leads that had clinical programming electrode that matched highest HFO power | 0
  DBS leads that had clinical programming row that matched highest HFO power | 2
  DBS leads that had clinical programming electrode that matched highest CFC | 0
  DBS leads that had clinical programming row that matched highest CFC | 5

2. Secondary Outcome: Number of DBS Leads With the Highest Side Effect Threshold at 3 Months That Were Consistent With Predictions Derived From LFPs After DBS Implant Procedure
Description: From all DBS leads (2 per patient):
  Local field potentials (LFPs) were measured intraoperatively during DBS implant. Features such as beta band power (10-30Hz), high-frequency oscillation power (200-400Hz, HFO), as well as the cross frequency coupling between beta band power and HFO (CFC) were extracted from the LFP recordings from all electrodes. Electrodes with the most beta band power, most HFOs, and most CFC were documented.
  At 3 month post-op visit, the stimulation electrode that produced the largest side effect threshold (any side effect) were documented, and were compared to the electrodes with the largest beta band, HFO, and CFC power documented from the intraoperative LFP measures.
Time Frame: LFPs were measured during DBS implant procedure, clinical programming were done at 3 month followup evaluation
Population: all patients with LFP data and who have gone through 3 month evaluation of side effect thresholds, each with bilateral implants
Measure: Count of Units; unit: DBS leads
Units Other Than Participants: DBS leads
Arm/Group | LFP Analyses From Patients With Bilateral Implants
Number analyzed (Participants) | 5
Number analyzed (DBS leads) | 10
DBS leads
  DBS leads that had highest side effect threshold contact predicted by HFO | 3
  DBS leads that had highest side effect threshold contact predicted by CFC | 3
  DBS leads that had highest side effect threshold contact predicted by beta-band power | 2

ADVERSE EVENTS:
Time Frame: surgery to 3 month post-surgery visit
Description: Both motor and non-motor side effect-induced adverse events were examined and reported.
Groups:
- LFP Recording Patients: All patients underwent STN DBS implants, 9/10 patients obtained LFP recordings during surgery. The 9 patients were then revisited for 3 month post-op followup.
Arm/Group | LFP Recording Patients
All-Cause Mortality (participants affected / at risk) | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 2/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LFP Recording Patients (N=10)
increased falls (Injury, poisoning and procedural complications) | 1 (1) — patient experienced increased gait issues and falls during Med off / stim on scenarios, the patient was withdrawn due to inability to tolerate off medication study assessments
cognitive impairment (Psychiatric disorders) | 1 (1) — patient became confused intraoperatively but surgical procedure was completed as planned. Due to persistent altered mental state, and MRI was ordered and showed bilateral edema

LIMITATIONS AND CAVEATS:
Medications/anesthesia could have an important effect on the LFP signal characteristic. For this reason local anesthesia should be used, as administration of anesthesia like propofol can wipe out or change the frequency spectrum of LFPs dramatically.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-09-29): https://cdn.clinicaltrials.gov/large-docs/02/NCT03630302/Prot_SAP_000.pdf